CLINICAL TRIAL: NCT03202407
Title: Effect of Non-calcium Phosphate Binders Versus Calcium Based Binders on Chronic Kidney Disease -Mineral and Bone Disorder in Children on Regular Hemodialysis
Brief Title: Hyperphosphatemia in Children With Chronic Kidney Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Ahmed, pediatrition, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEVELAMER
Record Dates: First submitted 2017-06-20; First posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — calcium acetate; Sevelamer

STUDY DESIGN:
Intervention Model Description: parallel group
Who Masked: Participant
Masking Description: single blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- calcium group (Placebo Comparator): will receive calcium-based phosphate binder (calcium carbonate ) 45-65 mg/kg orally divided 3 to 4 times/day for 3 months.
  all the following investigation will be done before and after consecutive 3 months of administration :
  * Complete blood count
  * Kidney function tests (serum urea and creatinine)
  * Serum total calcium level.
  * Serum phosphorus level.
  * Calcium × phosphorus product.
  * Serum parathormone level.
  * Serum alkaline phosphatase level.
  * Lipogram (Total cholesterol, High density lipoprotein, Low density lipoprotein and triglycerides).
  * Echocardiography regular follow up of serum phosphate , calcium and parathyroid hormone will be done every month for dose adjustment of the drug
  Interventions: Drug: Calcium acetate and sevelamer hydrochloride
- sevelamer group (Experimental): will receive the recommended daily dose of the Sevelamer hydrochloride phosphate binder 120-160 mg/kg orally 3 times per day for 3 months.
  all the following investigation will be done before and after consecutive 3 months of administration :
  * Complete blood count
  * Kidney function tests (serum urea and creatinine)
  * Serum total calcium level.
  * Serum phosphorus level.
  * Calcium × phosphorus product.
  * Serum parathormone level.
  * Serum alkaline phosphatase level.
  * Lipogram (Total cholesterol, High density lipoprotein, Low density lipoprotein and triglycerides).
  * Echocardiography regular follow up of serum phosphate , calcium and parathyroid hormone will be done every month for dose adjustment of the drug
  Interventions: Drug: Calcium acetate and sevelamer hydrochloride

INTERVENTIONS:
Drug: Calcium acetate and sevelamer hydrochloride — receive the conventional renal replacement therapy including calcium-based phosphate (calcium acetate) and active form of vitamin D for 3 months with regular follow up of serum phosphate ,calcium, parathyroid hormone and alkaline phosphate every month

SUMMARY:
"Chronic Kidney Disease-Mineral and Bone Disorder " is a systemic disorder of mineral and bone metabolism, due to chronic kidney disease that is manifested by either one or a combination of the following :

1. Abnormalities of calcium, phosphate, parathyroid hormone or vitamin D metabolism
2. Vascular and/or soft tissue calcification.
3. Abnormalities in bone turnover, metabolism, volume, linear growth or strength. According to glomerular filtration rate , Kidney Disease Improving Global Outcomesclassify chronic kidney disease into 5 stages,stage 5 also known as End Stage Renal disease is defined as glomerular filtration rate less than 15 ml/Min/1.73 m2, or the need for renal replacement therapy for survival The kidney plays a major role in phosphate homoeostasis. The kidneys excrete the total net amount of absorbed phosphate.Under normal physiological condition phosphate is freely filtered through the glomerulus. The majority (85-90%) of filtered phosphate undergoes tubular reabsorption primarily in proximal tubules.

Progressive renal insufficiency leads to hyperphosphatemia, hypocalcemia, and secondary hyperparathyroidism .

Hyperphosphatemia known as hidden killer in chronic kidney disease defined as an abnormally high serum phosphate concentration of >1.46 mmol/L (4.5 mg/dL). Its long term complications are renal osteodystrophy, hyperparathyroidism, and increased cardiovascular calcification leading to increased mortality and morbidity .

High serum phosphate can interact with calcium to precipitate calcium phosphate salts in non-skeletal tissues Calcification generally occurs in the blood vessels, heart valves, myocardium, and other soft tissues .

Cardiovascular calcification is probably the main reason for the high prevalence of cardiovascular diseases in chronic kidney disease patients Studies have shown that hyperphosphatemia is associated with increased vascular stiffening and arterial and valvular calcification This is postulated to be caused by elevated serum phosphorus promoting the transformation of vascular smooth muscle cells into an osteoblast phenotype that can mineralize These vascular calcification also lead to left ventricular hypertrophy by decreasing vascular compliance . Poor control of mineral metabolism also has been associated with functional and structural cardiac abnormalities Efforts to reduce morbidity and mortality associated with Chronic Kidney Disease-Mineral and Bone Disorder are therefore primarily directed at controlling hyperphosphatemia via diet, phosphorus binders, and dialysis

Dialysis alone is inadequate in assisting hemodialysis patients to obtain and maintain normal serum phosphate levels . So, other methods of achieving prescribed levels of serum phosphate in hemodialysis patients include the use of phosphate binders and phosphorus dietary restrictions.:

Phosphate binders have been approved by the Federal Drug Administration (FDA) for patients treated with maintenance dialysis, and calcium-containing salts are used worldwide not only for the control of hyperphosphatemia but also as a source of supplemental calcium. Several calcium salts are commercially available, including calcium carbonate, calcium acetate, and calcium citrate Sevelamer hydrochloride is a recently developed phosphate binder, which is a quaternary amine anion exchanger without calcium or aluminum. Sevelamer is effective in controlling hyperphosphatemia without increasing the calcium load in chronic hemodialysis patients In addition to its effects on serum phosphorous levels, sevelamer has been shown to decrease total serum cholesterol and low-density lipoprotein cholesterol and to increase high-density lipoprotein levels . These effects may offer additional benefits in reducing cardiovascular complications in patients with end-stage renal disease.

Controlling abnormal laboratory parameters such as calcium ,phosphate and parathyroid hormone as well as preventing the progression of extraskeletal calcification is considered a major component for prevention of the bone disease and other related morbidities and hopefully mortality in chronic kidney disease patients

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6 to 18 years
* With end stage renal disease on regular hemodialysis,
* With hyperphosphatemia (serum phosphorus > 4.5mg/dL ).
* Both genders will be included
* Given informed concent.

Exclusion Criteria:

* - Children < 6 years,
* Severe Gastrointestinal disorder,
* Known hypersensitivity to phosphate binders,
* Inability or rejection to give informed consent,
* Normal serum phosphate level.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
controlling of hyperphosphatemia | 3 months
  controlling abnormal laboratory parameters such as calcium, phosphate, and parathyroid hormone .
Cardiovascular complications | 3 months
  Preventing cardiovascular complication in children with chronic kidney disease